CLINICAL TRIAL: NCT03567044
Title: Outcomes and Immune Effects in Patients With Early Stage Breast Cancer Treated With Lumpectomy and Whole Breast Irradiation.
Brief Title: Immune Effects in Patients Treated With Whole Breast Irradiation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Shayna Showalter, MD, MD, Assistant Professor of Medicine, University of Virginia, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20476
Record Dates: First submitted 2018-03-13; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Collection (Experimental): Patients will be asked to have blood draws at specific time points during their whole breast irradiation.
  Interventions: Diagnostic Test: Blood Draw

INTERVENTIONS:
Diagnostic Test: Blood Draw — Eligible subjects will have blood draws at the following times: baseline, 1 week, 4 weeks, 8 weeks, 12 weeks, 24 weeks.

SUMMARY:
The purpose of this study is to obtain data to determine whether whole breast irradiation (WBI) differentially influences the frequency of components of innate and adaptive immunity and their relative functional activity, to assess the patient's quality of life (QOL) and to evaluate the cosmetic assessment of the breast on follow-up after WBI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide written informed consent and to comply with the study protocol as judges by the investigator.
* Patient has new diagnosis of breast cancer and has elected BCS and WBI. These patients must be consented prior to the start of WBI.
* For patients with invasive breast cancer sentinel node biopsy (SLNB) must be performed and confirm pathologic negative disease.
* Tumor size must be less than or equal to 3 cm.
* Patient is 45 years of age or older.
* Women of childbearing potential must agree to use adequate contraception prior to study entry and through the WBI treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Male patients
* Patients who are pregnant or nursing.
* Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the duration of the study or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Breast cancer that involves the skin or the chest wall.
* History of ipsilateral breast cancer treated with radiation therapy.
* Multicentric breast cancer in the ipsilateral breast as diagnosed by clinical exam, mammogram, ultrasound, or MRI
* Patients known to have a BRCA gene mutation. Genetic testing is not required.
* Patient with clinically positive nodal disease.
* Patient with proven nodal disease by either FNA, core biopsy or sentinel node biopsy.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Lymphopenia | Up to 6 months after treatment
  Incidence of lymphopenia
Cytokines | Up to 6 months after treatment
  Change in patient's number of cytokines

SECONDARY OUTCOMES:
Quality of Life | Up to 24 months after treatment
  Changes in Patient-Reported Quality of Life using the EORTC QLQ-C30
Cosmetic Changes | Up to 24 months after treatment
  Changes in physician reported cosmetic descriptions
Quality of Life | Up to 24 months after treatment
  Changes in Patient-Reported Quality of Life using the EORTC QLQ-BR23.
Cosmetic Changes | Up to 24 months after treatment
  Changes in patient reported cosmetic descriptions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No